CLINICAL TRIAL: NCT06330376
Title: Diaphragmatic Breathing Exercises for Post-COVID-19 Diaphragmatic Dysfunction (DD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-2022-30735
Record Dates: First submitted 2024-03-22; First posted 2024-03-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute Sequelae of COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: prospective randomized clinical study with 2 arms
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1 (Active Comparator): Participants randomized to usual care
  Interventions: Other: Usual care of traditional treatment
- arm 2 (Experimental): participants randomize to diaphragmatic breathing (DB) program
  Interventions: Other: Specific DB program/Diaphragmatic manipulation program

INTERVENTIONS:
Other: Usual care of traditional treatment — Usual care of traditional treatment which is PT and/or OT when indicated Followed by Pulmonary rehabilitation when indicated
  Arms: arm 1
Other: Specific DB program/Diaphragmatic manipulation program — 12 weeks of 2 sessions/week: one session will be remote and one in-person
  Arms: arm 2

SUMMARY:
Diaphragm is the principal muscle of inspiration. Diaphragmatic dysfunction is seen in many conditions including following intubation, lung disease, prolonged ventilation, neuromuscular disease, phrenic nerve injury. The possible mechanisms of diaphragmatic dysfunction in patients with COVID19 are critical illness myopathy, ventilator-induced diaphragm dysfunction, iatrogenic phrenic nerve injury particularly secondary to line placement, post-infectious inflammatory neuropathy of the phrenic nerve, or possibly direct neuromuscular involvement of the SARS- CoV-2 virus given expression of the angiotensin- converting enzyme 2 (ACE2) receptor in the peripheral nervous system and skeletal muscle. The use of diaphragmatic ultrasound has been widely used to assess diaphragmatic function is well known in patients following prolonged mechanical ventilation. Prolonged mechanical ventilation leads to contractile dysfunction of respiratory muscles, in particular the diaphragm, causing a so-called ventilator-induced diaphragm dysfunction. The latter is defined as a loss of diaphragm force-generating capacity specifically related to the use of mechanical ventilation. However, the use of diaphragmatic Ultrasound to assess its function in Long COVID patients has not been noted and is a gap in the work up of these patients.

The purpose of this study is to address Diaphragmatic Dysfunctional (DD) breathing seen in patients with Post-Acute Sequelae of COVID-19 (PASC), which results in shortness of breath/chest tightness and subsequent fatigue. Targeting shortness of breath and subsequent fatigue as a central symptom of PASC will alleviate long term sequelae for the patients with PASC. DD will be addressed by a unique intervention of physical therapy. The goal of this prospective randomized clinical study will be to evaluate the comparative treatment effect of DB on markers, specifically fatigue, dyspnea, 6 min walk test, depression/anxiety, and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 and above
* PCR or home kit positive 4 weeks prior to the development of the PASC symptoms
* new diagnosis of PASC (defined as new-onset symptoms of fatigue, shortness of breath, chest tightness or persistence of symptoms 4 weeks following a positive PCR test for COVID-19)
* patients did not need hospitalization of 5 days or more and did not need ICU admission via chart review or history taking.
* nose breathers as reported by patient at the time of screening by history taking
* symptoms should include shortness of breath/chest tightness/fatigue

Exclusion Criteria:

* pre-existing lung disease such as COPD, IPF, Asthma, Exercise induced Asthma, Lung cancer, or history of Lung transplant
* history of current smoking and pack years of 10
* history of coronary artery disease
* general anxiety disorder without changes in medication and dosage for treatment in the last 4 weeks.
* unable to have full range of motion of the shoulders
* stable dose of antidepressants prior to covid-19 infection
* Pregnant women/fetuses/neonates via self-report.
* non-English speakers
* patients with previously diagnosed severe cognitive deficits such as dementia, developmental defects, those with acute medical conditions, psychiatric disorders such as schizophrenia, mania, and psychosis, neurologic disorders such as stroke, Parkinson's disease and Multiple sclerosis
* unable to read
* Individual or group with a serious health condition for which there are no satisfactory standard treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | 6 months
  It is a simple test that requires no specialized equipment or advanced training for physicians and assesses the submaximal level of functional capacity of an individual while walking on a flat, hard surface in a period of 6 min. It is used to assess the response to a medical therapy, and in cardiac/pulmonary rehabilitation.

SECONDARY OUTCOMES:
PHQ9: Patient health questionnaire 9 | 6 months
  measures of depression, anxiety, and physical/mental/and social health, respectively, and will serve as covariates in our analysis.
GAD7: Generalized anxiety disorder 7-item | 6 months
  measures of depression, anxiety, and physical/mental/and social health, respectively, and will serve as covariates in our analysis.
PROMIS score: Patient-Reported Outcomes Measurement Information System | 6 months
  is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Administration of these scales is a standard of care in our post-COVID clinic.
QoL scale: Quality of life scale | 6 months
  measures of depression, anxiety, and physical/mental/and social health, respectively, and will serve as covariates in our analysis.
FACIT fatigue scale 's Fatigue score | 6 months
  Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (FACIT) FACIT fatigue scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (4 = not at all fatigued to 0 = very much fatigued) 18 The FACIT Fatigue Scale is one of many different FACIT scales that are part of a collection of health-related quality of life (HRQOL) questionnaires targeted to the management of chronic illness referred to as The FACIT Measurement System.
Modified Borg dyspnea scale | 6 months
  The Modified Borg Dyspnea Scale (MBS) is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administered during six-minute walk testing (6MWT).
RR; respiratory rate with 6 min walk test | 6 months
PR: pulse rate with 6 min walk test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Farha Ikramuddin, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States